CLINICAL TRIAL: NCT00989638
Title: A Multi Modality Surveillance Program for Women At High Risk for Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13073B
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women at high risk for breast cancer

SUMMARY:
The purpose of this study is to develop a coordinated, standardized screening program for the early detection of breast cancer in high-risk women. This would include Breast Mammography and Magnetic Resonance Imaging (MRI) examination of your breasts. The University of Chicago Department of Radiology is performing research to develop better ways of imaging the breast. The investigators would like to be able to reliably identify abnormal tissue and determine whether abnormal areas contain cancer without surgical procedures (i.e., a biopsy which involves removing breast tissue with a needle or surgical instrument). Annual mammography has already been recommended for the patient based on family history or personal history of cancer. In young women, dense breasts sometimes make it difficult to find abnormal changes on breast cancer screening (mammograms). MRI, in combination with mammography, may increase the rate of detection of early cancers. In addition, MRI can provide better images of breast tissue. The investigators hope to prove that combining multiple screening measures including biomarkers improves the chances that, if you have a small cancer or pre-cancer, it will be found early. This study will also evaluate quality of life measures during breast cancer screening and compare breast MRI and mammogram in a high-risk population. The investigators will establish a database of clinical characteristics, blood biomarkers and interventions that will be saved for future analysis and aid in the development of more effective screening in high-risk women. This research will also help us develop tools for studies in the future.

ELIGIBILITY:
Inclusion Criteria:

Each woman will meet one or more of the criteria below:

* Known BRCA1 or BRCA2 carrier (must be older than 21 years)
* Any mutation carrier in hereditary breast cancer susceptibility genes that is known to increase the risk for breast cancer (regardless of age). Some examples of these would include TP53, PTEN, BRCA1 and BRCA2, CHEK2, ATM, and CDH1 and other identified genetic markers conferring greater than 2.5 fold increased breast cancer risk in a polygenic model.
* For women who chose not to have genetic testing or test negative, probability of being a BRCA1 or BRCA2 carrier of 20% or greater based on BRCAPRO analysis or ≥ 25% risk of being a mutation carrier by any Genetic model such as Couch, Myriad, BODICEA, in addition to a lifetime breast cancer risk >=20% by CARE, Tyler Cuzick, or Claus model
* Personal history of breast cancer before age 35 years and no evidence of disease recurrence for at least two years.
* Any woman of African ancestry whose 1st degree relative (mother or sister) or 2nd degree relative (aunt, grandmother) if paternal lineage suspected diagnosed with breast cancer under age 40, regardless of risk model calculation
* Have a personal history of ductal carcinoma in situ (DCIS) diagnosed at or before age 35 AND a first degree relative who had been diagnosed with breast cancer before age 50 OR has a first degree relative diagnosed with ovarian cancer at any age
* Any female cancer survivor who received chest irradiation before age 30 for any disease including Hodgkin's, a sarcoma, neuroblastoma, or other medical condition.

In addition to meeting one of the above criteria, women must meet all of the following:

* willing to travel to University of Chicago Medical Center for imaging studies as well as any necessary follow-up procedures.
* have at least one breast that has not been irradiated for cancer
* be at least 25 years of age or at least 5 years younger than the first case of breast cancer diagnosis in the family. (This applies only to high risk women who are not BRCA1 or BRCA2 mutation carriers)
* be able to give informed consent

Exclusion Criteria:

Women will be excluded if they meet one of the following:

* active cancer at the time of enrollment. A prior history of breast cancer is permitted if the subject has completed chemotherapy and is considered disease-free at the time of enrollment.
* current pregnancy or plans for pregnancy within two years of enrollment
* presence of a pacemaker or any other metallic foreign objects in their body that interferes with an MRI
* breast surgery within two weeks of study entry
* previous bilateral mastectomy (prophylactic or therapeutic)
* history of kidney disease or abnormal kidney tests
* Women who test negative in a family with identifiable BRCA mutations are ineligible regardless of risk calculation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women at high risk for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2004-06-23 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Creation of registry of women undergoing intensive surveillance for the early detection of breast cancer in high-risk women | Until enrollment is complete
Impact of intensive breast cancer screening on patient reported outcomes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo Olopade, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Guindalini RSC, Zheng Y, Abe H, Whitaker K, Yoshimatsu TF, Walsh T, Schacht D, Kulkarni K, Sheth D, Verp MS, Bradbury AR, Churpek J, Obeid E, Mueller J, Khramtsova G, Liu F, Raoul A, Cao H, Romero IL, Hong S, Livingston R, Jaskowiak N, Wang X, Debiasi M, Pritchard CC, King MC, Karczmar G, Newstead GM, Huo D, Olopade OI. Intensive Surveillance with Biannual Dynamic Contrast-Enhanced Magnetic Resonance Imaging Downstages Breast Cancer in BRCA1 Mutation Carriers. Clin Cancer Res. 2019 Mar 15;25(6):1786-1794. doi: 10.1158/1078-0432.CCR-18-0200. Epub 2018 Aug 28. PMID 30154229